CLINICAL TRIAL: NCT00142623
Title: Reducing ETS Exposure of Pregnant Women and Newborns
Brief Title: Tailored Videos to Reduce Tobacco Smoke Exposure Among Pregnant Women and Newborns
Acronym: ETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Thomas M. Lasater, PhD, Brown University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 249; R01HL070947 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Use of five tailored "take-home" DVDs aimed at reducing exposure to ETS
  Interventions: Behavioral: Tailored DVDs
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Tailored DVDs — Five DVDs aimed at reducing exposure to ETS
  Arms: 1

SUMMARY:
The purpose of this study is to develop and evaluate the efficacy of five tailored DVDs in reducing exposure to environmental tobacco smoke (ETS) among low income pregnant/postpartum women.

DETAILED DESCRIPTION:
BACKGROUND:

The Healthy People 2010 Objectives address the importance of smoking cessation during pregnancy and the importance of reducing ETS exposure among children and adults. This study will use a new combination of existing technologies to maximize the appropriateness of prenatal and postpartum education concerning ETS exposure in an innovative, inexpensive, and widely applicable approach. The use of tailored DVDs is practical, feasible, and inexpensive enough to be attractive to clinics serving low-income and minority women. A large number of video segments will be produced utilizing live actors, animation, and word slates. About 10 segments will be computer-selected for the videos for each woman based on her responses to four self-assessments. No studies to date have included multiple doses of tailored video education, or used DVDs in this way.

DESIGN NARRATIVE:

This two-arm randomized study is designed to develop and evaluate the efficacy of five tailored DVDs in reducing exposure to ETS among low-income pregnant/postpartum women. The overall purposes of the study are 1) to develop an innovative intervention (tailored "take-home" DVDs) to help pregnant women maximize their pregnancy outcome and their new infant's health through reduction in exposure to ETS and 2) to study the feasibility and efficacy of this intervention compared with a usual care group. This innovative technology will be field tested in collaboration with six prenatal clinics that serve primarily low-income, African American, Latina, and minority women to address two specific aims. Specific aim 1: To test the efficacy of tailored video (TV) versus usual care (UC) approaches in terms of reducing the ETS exposure among fetuses of nonsmoking, low-income women during pregnancy (assessed at 34 weeks gestation using saliva cotinine concentration and ETS self-report) and among infants (as measured by saliva cotinine concentration and mothers' self-reports at 6 months postpartum). Specific aim 2: To test the efficacy of TV versus UC approaches in terms of reducing the exposure of the fetuses of low-income, smoking women to tobacco smoke during pregnancy (assessed at 34 weeks gestation using saliva cotinine concentrations of the pregnant women and smoking and ETS self-reports) and to their infants (as measured by saliva cotinine concentration from the infant at 6 months postpartum and self-reports of infant exposure by the new mothers). Because of the lack of data on reducing ETS exposure amongst low-income and minority women, intensive formative and extensive process evaluation components are included.

ELIGIBILITY:
Inclusion Criteria:

* Women who attend their first prenatal visit by 16 weeks gestation
* Women exposed to tobacco smoke daily

Exclusion Criteria:

* Women expecting complications or multiple births

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Saliva cotinine concentration of mother | Measured at 34 weeks gestation
ETS self-report | Measured at 34 weeks gestation and 6 months postpartum
ETS exposure of infant by self-report of mother | Measured at 6 months postpartum
Salvia cotinine concentration of infant | Measured at 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Lasater, PhD, Principal Investigator — Brown University; Patricia M. Risica, DrPH, Principal Investigator — Brown University; Maureen Phipps, MD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States